CLINICAL TRIAL: NCT06672198
Title: "Evaluation of Elective Cesarean Surgery Within the Scope of ERAC Protocol: Where Are We in Türkiye"
Brief Title: ERAC Protocol in Elective Cesarean Surgery
Acronym: Erac
Status: Completed | Type: Observational
Sponsor: Gonca Karatas Baran (Other)
Responsible Party: Sponsor-Investigator, Gonca Karatas Baran, Dr Nurse, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Organization: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Other Study IDs: gkbaran
Record Dates: First submitted 2024-10-25; First posted 2024-11-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cesrean Delivery; Enhanced Recovery After Surgery
Keywords: Cesarean section; Enhanced recovery after surgery; Perioperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- cesarean delivery: women undergoing elective caesarean section
  Interventions: Procedure: ERAC protocol

INTERVENTIONS:
Procedure: ERAC protocol — our study aimed to evaluate pre-peri-post operative practices in women who underwent elective cesarean section (CS) according to the ERAC protocol. In this context, this study aimed to describe the implementation status of the recommendations regarding the ERAC protocol in CS operations, to identify the missing aspects of the ERAC protocol and to raise awareness about its benefits.

SUMMARY:
This descriptive prospective study was conducted between 01/12/2021-01/09/2022. The sample of the study consisted of 333 women who underwent elective cesarean section (CS). Nurse observation form, anesthesia follow-up form, patient file and verbal expressions of women were used to collect data. Number, percentage, mean and standard deviation were used as descriptive statistics.

DETAILED DESCRIPTION:
A descriptive prospective study was conducted in the Gynecology and Obstetrics branch hospital between 01/12/2021-01/09/2022. The universe of the study consisted of pregnant women who underwent elective CS in the relevant hospital. The study sample consisted of 333 patients who underwent elective CS with the sample calculation method when the universe was known (N: Number of individuals in the population (2500), p: Incidence of the investigated event (0.5), q: Incidence of the examined event (0.5), t: Certain theoretical value found in the "t" table at the degree of freedom and the detected error level (1.96), d: Sensitivity to be made according to the incidence of the event (0.05), 0.95 confidence interval, 0.05 margin of error).

The period of the study group was followed from hospitalization to discharge. The data collection form prepared by scanning the literatüre1-6 was used to collect the research data. The data collection form consisted of two parts. In the first part, there were questions about the socio-demographic and obstetric characteristics of the participant, and in the second part, questions about the components of the ERAC protocol. Nurse observation form, anesthesia follow-up form, patient file and verbal expressions of women were used to collect data. In the research, data related to health practices were taken from the file and recorded. Inclusion criteria; women who agreed to participate in the study, who were hospitalized in the CS, and who had elective CS surgery. Women who did not have elective CS and did not accept participation in the study are exclusion criteria.

Ethics committee approval was obtained from the clinical research ethics committee for the study and informed consent was obtained from the participants.

The analysis of the data was done in computer environment with SPSS (Statistical Package for the Social Sciences) 20.0 ready-made statistical program. In the evaluation of the data; number, percentage, mean and standard deviation were used as descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria; women who agreed to participate in the study, who were hospitalized in the CS, and who had elective CS surgery

Exclusion Criteria:

* Women who did not have elective CS and did not accept participation in the study are exclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women who were hospitalized in the CS.
Study Population: women who had elective CS surgery in the XX hospital
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Preoperative applications | from december 2021 to september 2022
  Sedative premedication Yes No
Preoperative information | from december 2021 to september 2022
  Preoperative IV fluid ......cc
Preoperative information , | from december 2021 to september 2022
  Preoperative LMWH aplication Yes No
Preoperative information | from december 2021 to september 2022
  Preoperative antibiotic prophylaxis Yes No
Preoperative information | from december 2021 to september 2022
  Bowel preparation Yes No
Preoperative information | from december 2021 to september 2022
  Skin cleansing with chlorhexidine Yes No
Preoperative information | from december 2021 to september 2022
  ASA classification I, II, III
Preoperative information | from december 2021 to september 2022
  Solid food restriction period (hour)....hour
Preoperative information | from december 2021 to september 2022
  Liquid food restriction period (hour)....hour
Intraoperative applications | from december 2021 to september 2022
  Type of anesthesia General, spinal
Intraoperative applications | from december 2021 to september 2022
  NG cathetere application yes No
Intraoperative applications | from december 2021 to september 2022
  Urinary catheterization application Yes No
Intraoperative applications | from december 2021 to september 2022
  Drain application Yes No
Intraoperative applications | from december 2021 to september 2022
  Epidural analgesia administration Yes No
Intraoperative applications | from december 2021 to september 2022
  Antiemetic agent administration Yes No
Intraoperative applications | from december 2021 to september 2022
  Intraoperative IV fluid amount (cc)......cc
Intraoperative applications | from december 2021 to september 2022
  Incision length (cm).......cm
Postoperative applications | from december 2021 to september 2022
  Nausea Yes No
Postoperative applications | from december 2021 to september 2022
  Heating with a heater Yes No
Postoperative applications | from december 2021 to september 2022
  Pain score (VAS)1-10
Postoperative applications | from december 2021 to september 2022
  Analgesic administration Yes No
Postoperative applications | from december 2021 to september 2022
  Type of analgesic ........
Postoperative applications | from december 2021 to september 2022
  Posoperative LMWH application Yes No
Postoperative applications | from december 2021 to september 2022
  Gum chewing app yes No
Postoperative applications | from december 2021 to september 2022
  Status of providing discharge training Yes No
Postoperative applications | from december 2021 to september 2022
  Information on control Yes No
Postoperative applications | from december 2021 to september 2022
  Principle time breastfeeding (minute).......minute
Postoperative applications | from december 2021 to september 2022
  Time to postoperative gas release (hour)........hour
Postoperative applications | from december 2021 to september 2022
  Time to postoperative stool output (hour).......hour
Postoperative applications | from december 2021 to september 2022
  Time to mobilization (hour)...........hour later
Postoperative applications | from december 2021 to september 2022
  Time to urinary catheter removal (hour)..........hour kater
Postoperative applications | from december 2021 to september 2022
  Time to oral initiation (hour)........hour
Postoperative applications | from december 2021 to september 2022
  Hospitalization time (hour)........hour

SECONDARY OUTCOMES:
socio-demographic characteristics. | from december 2021 to september 2022
  data on socio-demographic characteristics

CONTACTS AND LOCATIONS:
Overall Officials: gonca Karataş Baran, phd, Principal Investigator — Etlik Zübeyde Hanım Maternity and Women's Health Teaching and Research Hospital
Locations (1):
- Etlik Zübeyde Hanım Maternity and Women's Health Teaching and Research Hospital, Ankara, yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided